CLINICAL TRIAL: NCT06324162
Title: Does the Pain Experienced During Orthodontic Treatment and Bracket Removal Depend on the Architecture of the Bracket? A Comparative Study of Two Bracket Systems and Two Debonding Methods
Brief Title: Does the Pain Experienced During Orthodontic Treatment and Bracket Removal Depend on the Architecture of the Bracket?
Acronym: Debonding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Piotr Fudalej (Other)
Responsible Party: Sponsor-Investigator, Piotr Fudalej, Prof. dr hab., Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JagiellonianU Gibas-Stanek
Record Dates: First submitted 2024-03-03; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Debonding; Orthodontic Brackets
Keywords: orthodontic brackets; pain measurement; dental debonding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2-slot brackets (Experimental): 50 patients treated with 2-slot brackets.
  Interventions: Device: bracket removal pliers, LODI
- Twin brackets (Experimental): 50 patients treated with traditional twin brackets.
  Interventions: Device: bracket removal pliers, LODI

INTERVENTIONS:
Device: bracket removal pliers, LODI — Brackets on the right side of both dental arches were debonded using the lift-off debonding instrument (LODI), while on the left side, the bracket removal pliers (BRP). The residual adhesive was removed through two methods (manual in the upper arch and rotary in the lower). The same scale was employed to assess pain levels during brackets and adhesive removal.
  Other Names: adhesive removal pliers, tungsten bur

SUMMARY:
The present research aimed to thoroughly investigate the impact of bracket architecture on pain perception during active treatment, debonding, and adhesive removal.

DETAILED DESCRIPTION:
100 consecutive patients who completed treatment with one of two bracket systems (2-slot brackets with integral base or conventional twin brackets with foil mesh) were included in this prospective clinical trial. Prior to the removal of brackets, participants were asked to evaluate the level of pain encountered throughout their orthodontic treatment with the fixed appliances, utilizing a 0-10 numerical rating scale, and to indicate the main cause of pain. Subsequently, brackets on the right side of both dental arches were debonded using the lift-off debonding instrument (LODI), while on the left side, the bracket removal pliers (BRP). The residual adhesive was removed through two methods (manual in the upper arch and rotary in the lower). The same scale was employed to assess pain levels during brackets and adhesive removal.

ELIGIBILITY:
Inclusion Criteria:

* fixed appliance in both dental arches
* brackets bonded using the Transbond XT adhesive system (3M Unitek, St. Paul, USA) following the manufacturer's instructions

Exclusion Criteria:

* periodontal disease
* restorations or caries on buccal surfaces of the teeth,
* consumption of analgesics within eight hours preceding the debonding appointment

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Pain during active treatment | On the day of debondig (at the end of active treatment).
  Numerical Rating Scale (0-10) was used to assess pain level during active treatment.
Pain during brackets removal | On the day of debondig (after debonding of each single bracket).
  Numerical Rating Scale (0-10) was used to assess pain during brackets debonding.
Pain on adhesive removal | On the day of debondig (after adhesive removal in each quadrant).
  Numerical Rating Scale (0-10) was used to assess pain during adhesive removal.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Fudalej, Prof., Study Director — Department of Orthodontics, Jagiellonian University Medical College
Locations (1):
- Jagiellonian University Collegium Medicum, Krakow, Poland

REFERENCES:
- [Derived] Gibas-Stanek M, Fudalej P. Does the pain experienced during orthodontic treatment and bracket removal depend on the architecture of the bracket or debonding method? Eur J Orthod. 2024 Dec 4;47(1):cjae073. doi: 10.1093/ejo/cjae073. PMID 39665482